CLINICAL TRIAL: NCT04425382
Title: Efficacy and Safety of Darunavir/Cobicistat vs. Lopinavir/Ritonavir in the Management of Patients With COVID-19 Pneumonia in Qatar
Brief Title: Darunavir/Cobicistat vs. Lopinavir/Ritonavir in COVID-19 Pneumonia in Qatar
Acronym: DOLCI
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-05-069
Record Dates: First submitted 2020-05-21; First posted 2020-06-11 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus; COVID; Pneumonia
MeSH Terms: conditions — Coronavirus Infections; Pneumonia | interventions — cobicistat mixture with darunavir; Lopinavir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Darunavir/Cobicistat: Patients received Darunavir/Cobicistat (Rezolsta®) as part of the treatment regimen for COVID-19 pneumonia
  Interventions: Drug: Darunavir/Cobicistat
- Lopinavir/Ritonavir: Patient received Lopinavir/Ritonavir (Kaletra®) as part of the treatment regimen for COVID-19 pneumonia
  Interventions: Drug: Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Darunavir/Cobicistat — Darunavir/Cobicistat (800mg/150mg) 1 tablet PO once daily
  Groups: Darunavir/Cobicistat
Drug: Lopinavir/Ritonavir — Lopinavir/Ritonavir (200mg/50mg) 2 tablets PO twice daily
  Groups: Lopinavir/Ritonavir

SUMMARY:
Coronavirus Disease 2019 (COVID-19) is a disease caused by the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) virus. It was first isolated in Wuhan, China in December 2019 and then rapidly spread to the rest of the world posing a severe threat to global health.

Many therapeutics have been investigated for the treatment of this disease with inconclusive outcomes. Protease inhibitors are one of the proposed agents, but their use is limited to their significant drug interactions and side effects.

The aim of this study is to compare the efficacy and safety outcomes of Darunavir/Cobicistat versus Lopinavir /Ritonavir in the treatment of patients with COVID-19 pneumonia in Qatar.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years of age
* Laboratory confirmed 2019-nCoV infection as determined by the PCR of the nasopharyngeal/oropharyngeal swab.
* Radiologically confirmed pneumonia (Based on the chest x-ray or CT scan imaging).
* Have received either Darunavir/Cobicistat or Lopinavir/Ritonavir as part of the treatment regimen for COVID-19 pneumonia

Exclusion Criteria:

* No exclusion criteria will be applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient who were admitted to HMC hospitals with laboratory confirmed 2019-nCoV infection who meet the inclusion criteria during the review period will be included.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Time to Clinical Improvement and/or Virological Clearance (Composite Endpoint) | Up to 90 days
  * Clinical Improvement is defined as the time to normalization of fever (defined as temperature <37.8 oC for 72 hours) and/or resolution of baseline sign/symptoms, without the need for symptomatic treatment
  * Virological clearance is defined as the time to two consecutive negative COVID-19 PCR samples

SECONDARY OUTCOMES:
Percentage of Virological Clearance | At day 14, day 21, and day 28.
  o Defined as two consecutive negative COVID-19 PCR samples
Percentage of Clinical Deterioration | Up to 28 days
  o Defined as the need for respiratory support, vasopressor use, or corticosteroids/immunomodulation therapy
Incidence of Adverse Events | Up to 28 days
Length of Hospital Stay | Up to 90 days
All-cause Mortality | At 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Eman Elmekaty, PharmD, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elmekaty EZI, Alibrahim R, Hassanin R, Eltaib S, Elsayed A, Rustom F, Mohamed Ibrahim MI, Abu Khattab M, Al Soub H, Al Maslamani M, Al-Khal A. Darunavir-cobicistat versus lopinavir-ritonavir in the treatment of COVID-19 infection (DOLCI): A multicenter observational study. PLoS One. 2022 May 4;17(5):e0267884. doi: 10.1371/journal.pone.0267884. eCollection 2022. PMID 35507606